CLINICAL TRIAL: NCT00217594
Title: A Pilot Study of Alemtuzumab (Campath[R]) in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: A Pilot Study of Alemtuzumab (Campath[R]) in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050206; 05-H-0206; NCT00123721 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2017-10-17

CONDITIONS: Myelodysplastic Syndromes
Keywords: Immunosuppression; T Cells; Hematopoiesis; Anti-CD52; Monoclonal Antibody Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alemtuzumab (Experimental): Patients received a 1-mg test dose of alemtuzumab, and the following day, alemtuzumab was administered at 10 mg/dose intravenously for 10 days
  Interventions: Drug: Alemtuzumab (Campath)

INTERVENTIONS:
Drug: Alemtuzumab (Campath)

SUMMARY:
This study will evaluate the safety and effectiveness of a genetically engineered antibody, alemtuzumab (Campath[R]) on patients with myelodysplastic syndrome. MDS is made up of malignant stem cell disorders that can mean low levels of red blood cells-that is, anemia-and low counts of white blood cells and platelets. Patients with MDS are at risk for infection, spontaneous bleeding, and possible progression to leukemia, a cancer of bone marrow. Although bone marrow can produce some blood cells, patients with MDS experience a decrease in production of blood cells. Alemtuzumab recognizes specific types of white cells called lymphocytes and destroys them. This study will examine not only the usefulness of the medication but also the side effects in patients with MDS.

Patients ages 18 to 72 who have MDS that requires transfusions and who do not have HIV or a life expectancy of less than 6 months may be eligible for this study. Screening tests include a complete physical examination and medical history. There will be a collection of about 8 tablespoons of blood for analysis of blood counts as well as liver, kidney, and thyroid function; a pregnancy test; an electrocardiogram (EKG) to measure electrical activity of the heartbeat; an echocardiogram (ECHO), which uses sound waves to evaluate heart function; wearing of a Holter monitor for 24 hours while the electrical activity of the heart is recorded; and a bone marrow biopsy. Patients should not receive any vaccines when taking alemtuzumab or for at least 12 months after the last dose. In addition, patients should not take the herbal supplements Echinacea purpurea or Usnea 2 weeks before beginning the study and during it.

For the study, all patients will receive a test dose of 1 mg of alemtuzumab infused into a vein during the course of 1 hour. If the dose is tolerated, the medication will be given at 10 mg doses into the vein for 10 days, as an infusion of 2 hours. Blood samples of 2 tablespoons will be taken daily, and vital signs will be measured daily. The ECHO and 24-hour Holter monitoring will be repeated after patients receive the last dose of the medication. Because suppression of the immune system results from a decrease in white cells that fight infections, patients will take medications to protect them against infections and to treat them if infections occur. If needed, patients will receive blood transfusions for their MDS. Side effects of alemtuzumab involve a temporarily significant lowering of the number of red blood cells, white cells, and platelets. Side effects of the infusion can be rigidity, or stiffness, and fever, as well as risks of infections resulting from the decrease of white blood cells. Blood counts and reactions to all procedures will be carefully monitored throughout the study. After patients receive the last dose of alemtuzumab, they will have follow-up by their referring doctor or at NIH. They must be able to return to NIH after 1 month, 3 months, 6 months, and annually for 5 years after the study. At follow-up visits, there will be blood tests to reevaluate blood counts and test for the presence of viruses. Blood tests will be done weekly for the first 3 months after patients have completed taking alemtuzumab, every other week until 6 months, and then annually for 5 years. There will also be a repeat ECHO at the 3-month visit, and a repeat bone marrow biopsy at the 5-month and 12-month follow-up visits, and as needed after that.

This study may or may not have a direct benefit for participants. For some, the antibody may improve blood counts and decrease the need for transfusions. Knowledge gained in the study may help people in the future.

DETAILED DESCRIPTION:
Many bone marrow failure syndromes in humans are now recognized to result from immunological mechanisms. These diseases include aplastic anemia, pure red cell aplasia, and some types of myelodysplasia. Patients with these conditions, who may suffer variable degrees of anemia, leukopenia, and thrombocytopenia, alone or in combination, have been shown to respond to a wide variety of immunosuppressive agents, ranging from corticosteroids to cyclosporine (CsA) and horse antithymocyte globulin (h-ATG). However, non-response and relapse continues to be a problem. Why some patients do not respond initially or others respond and then relapse is unclear. Autoreactive T cells may be resistant to the effect of h-ATG/CsA (non-responders), while in others, residual autoreactive T cells expand post-treatment leading to hematopoietic stem cell destruction and recurrent pancytopenia (relapse). Therefore, novel, less toxic immunosuppressive regimens that increase response rates and hematologic recovery and decrease relapse rates are needed.

One such novel therapy, alemtuzumab (Campath[R]) is a humanized IgG1 monoclonal antibody directed against the CD52 protein, which is highly expressed on all lymphoid cells and monocytes. Alemtuzumab (Campath[R]), produces profound and persistent lymphopenia, affecting predominantly the CD4+ T cell subset. This property has made it attractive in the treatment of a wide range of diseases including rheumatoid arthritis, multiple sclerosis, ocular inflammatory disease, lymphoid malignancies, organ allograft rejection, and in conditioning regimens in stem cell transplantation to prevent graft failure and graft-versus-host disease.

We therefore propose a non-randomized, off label, pilot, Phase I/II study of alemtuzumab (Campath) in MDS patients who are likely to respond to immunosuppression.

Primary endpoints will be changes in peripheral blood counts (platelets, absolute neutrophil count, reticulocyte count, hemoglobin). Secondary endpoints (in transfusion-dependent patients) include improvement in the transfusion requirements (measured as decrease in the number of transfusion administered on as needed basis), duration of response, late effects of treatment, relapse and survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. MDS with WHO classification of RA, RARS, RCMD-RS, RCUD, and RCMD and RAEB-1 (all subtypes of MDS with the exception of RAEB 2, CMML, and MDS/MPN overlap)
  2. Anemia requiring transfusion support with at least one unit of packed red blood cells per month for greater than or equal to 2 months

     OR

     Anemia (hemoglobin less than 9 or a reticulocyte count less than 60,000)

     OR

     thrombocytopenia (platelet count less than 50000/ul)

     OR

     neutropenia (absolute neutrophil count less than 500/ul).
  3. Off all other treatments for MDS (except filgrastim (G-CSF), erythropoietin, and transfusion support and related medications) for at least four weeks. Filgrastim (G-CSF) can be used before, during and after the protocol treatment for patients with documented neutropenia (less than 500/Ul) as long as they meet the criteria for anemia and/or thrombocytopenia as stated above.
  4. Ages 18-72 (inclusive)

EXCLUSION CRITERIA:

1. Chronic myelomonocytic leukemia (CMML), MDS/MPN overlap, WHO RAEB-2
2. Secondary MDS
3. Failure to respond to prior therapy with ATG or ATG/CsA
4. Prior therapy with combination chemotherapy
5. Transformation to acute leukemia (FAB sub-group RAEB-T, i.e., greater than 20% blasts in marrow aspirate)
6. Failure to discontinue the herbal supplements Echinacea purpurea or Usnea barbata (Old Man's Beard) within 2 weeks of enrollment.
7. Active infection not adequately responding to appropriate therapy
8. HIV positive patients
9. Active malignant disease (excluding non-melanoma skin carcinoma)
10. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy or that death within 7-10 days is likely.
11. Life expectancy less than 6 months
12. Low predicted probability of response
13. Previous hypersensitivity to alemtuzumab (Campath[R]) or its components
14. Current pregnancy, or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential
15. Not able to understand the investigational nature of the study or give informed consent

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07-21; Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hourigan, BMBCh, Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nydegger UE. Suppressive and substitutive immunotherapy: an essay with a review of recent literature. Immunol Lett. 1985;9(4):185-90. doi: 10.1016/0165-2478(85)90031-8. No abstract available. PMID 3888832
- [Background] Tichelli A, Gratwohl A, Wuersch A, Nissen C, Speck B. Antilymphocyte globulin for myelodysplastic syndrome. Br J Haematol. 1988 Jan;68(1):139-40. doi: 10.1111/j.1365-2141.1988.tb04194.x. No abstract available. PMID 3345291
- [Background] Biesma DH, van den Tweel JG, Verdonck LF. Immunosuppressive therapy for hypoplastic myelodysplastic syndrome. Cancer. 1997 Apr 15;79(8):1548-51. doi: 10.1002/(sici)1097-0142(19970415)79:83.0.co;2-y. PMID 9118037
- [Result] Sloand EM, Olnes MJ, Shenoy A, Weinstein B, Boss C, Loeliger K, Wu CO, More K, Barrett AJ, Scheinberg P, Young NS. Alemtuzumab treatment of intermediate-1 myelodysplasia patients is associated with sustained improvement in blood counts and cytogenetic remissions. J Clin Oncol. 2010 Dec 10;28(35):5166-73. doi: 10.1200/JCO.2010.29.7010. Epub 2010 Nov 1. PMID 21041705
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] Hosokawa K, Kajigaya S, Feng X, Desierto MJ, Fernandez Ibanez MD, Rios O, Weinstein B, Scheinberg P, Townsley DM, Young NS. A plasma microRNA signature as a biomarker for acquired aplastic anemia. Haematologica. 2017 Jan;102(1):69-78. doi: 10.3324/haematol.2016.151076. Epub 2016 Sep 22. PMID 27658437

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 40 enrolled subjects, only 31 subjects were evaluable.
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 57 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 24
  Race/Ethnicity: African American | 2
  Race/Ethnicity: Asian | 2
  Race/Ethnicity: Hispanic | 3

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment - Hematologic Improvement or Complete Response
Description: Response to treatment at 3 months after the first dose of alemtuzumab. The parameters for hematologic improvement (HI) and complete response (CR) were defined according to the International Working Group (IWG) criteria. The IWG criteria for HI define specific responses of cytopenias in the 3 hematopoietic lineages: erythroid (HI-E), platelet (HI-P), and neutrophil (HI-N).7 The HIs are measured in patients with pretreatment abnormal values: hemoglobin level less than 110 g/L (11 g/dL) or RBC-transfusion dependence, platelet count less than 100 × 109/L or platelet-transfusion dependence, absolute neutrophil count (ANC) less than 1.0 × 109/L.
  The parameters for CR include less than 5% marrow blasts without evidence of dysplasia and normalization of peripheral blood counts, including a hemoglobin level of 110 g/L (11 g/dL) or more (in patients not receiving erythropoietin or transfusions), a neutrophil count of 1.5 × 109/L or more, and a platelet count of 100 × 109/L.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 31
Participants | 21

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 15/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab (N=31)
Bacterial pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile diarrhea (Infections and infestations) | 2
Neutropenic fever (Infections and infestations) | 3
Non-neutropenic fever (Infections and infestations) | 2
Shingles (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
URI symptoms (Infections and infestations) | 1
Hypotension (Injury, poisoning and procedural complications) | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1
Molluscum contagiosum skin lesion (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab (N=31)
Hypertension (Cardiac disorders) | 1
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
Stiffness (General disorders) | 1
Facial flushing (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infusion reaction (Injury, poisoning and procedural complications) | 23
Orchitis (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Upper respiratory tract (Infections and infestations) | 9
Mycobacterium chelonae (Infections and infestations) | 1
Hand swelling (Blood and lymphatic system disorders) | 1
Decreased phosphate (Metabolism and nutrition disorders) | 1
Elevated AST, ALT (Metabolism and nutrition disorders) | 8
Elevated LDH (Metabolism and nutrition disorders) | 1
Elevated creatinine (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (General disorders) | 2
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3
Neuropathic (Nervous system disorders) | 1
Darkened urine (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT00217594/Prot_SAP_000.pdf